CLINICAL TRIAL: NCT05856500
Title: A Prospective Open Controlled Study of Creatine Combined With Curcumin in the Intervention of Early Cachexia in Upper Gastrointestinal Tumors
Brief Title: A Study of Creatine Combined With Curcumin in the Intervention of Early Cachexia in Upper Gastrointestinal Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-223-02
Record Dates: First submitted 2022-12-05; First posted 2023-05-12 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-12

CONDITIONS: Stage IV Gastric Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage III Esophageal Cancer; Stage IV Esophageal Cancer
Keywords: Creatine; Cur-cumin; Early Cachexia
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Cachexia | interventions — Curcumin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- basic nutrition (Placebo Comparator): basic nutrition treatment, energy 30-35 kcal/kg, protein 1.0-2.0 g/kg, total nutrition and/or whey protein oral nutrition supplement or tube feeding enteral nutrition supplement if diet deficiency;
  Interventions: Dietary Supplement: basic nutrition
- oral supplement of creatine and curcumin (Experimental): On the basis of basic nutrition in group A, creatine 5g/d and curcumin 4g/d are orally added, and the intervention time is 1 month.
  Interventions: Dietary Supplement: oral supplement of creatine and curcumin

INTERVENTIONS:
Dietary Supplement: basic nutrition — An adequate supply of energy and protein in diet, oral nutrition supplement or tube feeding enteral nutrition supplement when diet is deficient.
  Arms: basic nutrition
Dietary Supplement: oral supplement of creatine and curcumin — Creatine and curcumin are orally added other than basic nutrition treatment.
  Arms: oral supplement of creatine and curcumin

SUMMARY:
Cachexia is a common complication of various advanced malignant tumors, which seriously affects the quality of life and survival time of patients. In view of the clinical problem of non-nutritional response in patients with cachexia, the investigators plan to carry out a clinical case-control study on the intervention of creatine combined with curcumin in participants with cachexia. On the whole, the investigators limited the study subjects to upper digestive tract tumors and diagnosed participants with early cachexia. The main purpose of this study is to determine whether the combination of the two can play a positive and stable role in inhibiting the inflammation of cachexia and improving metabolic status, so that basic nutrition can play a role, in order to reduce the level of skeletal muscle consumption, maintain weight, improve quality of life, save medical costs and extend survival time.

DETAILED DESCRIPTION:
This is a prospective open controlled study. The intervention is targeted at participants with early cachexia in upper gastrointestinal tumors.Both control group and intervention group receive basic nutritional support. On the basis of this, the intervention group will be given creatine and curcumin orally.The purpose is to investigate whether creatine combined with curcumin can improve the inflammatory and the nutritional state, correct the disorder of nutrient metabolism and improve the prognosis of participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced tumors of the upper digestive tract with untreatable or postoperative recurrence of esophageal and gastric cancer III-IV
* Meet the diagnostic criteria of early cachexia (anorexia and metabolic changes, involuntary body mass reduction ≤5% within 6 months)
* Radiotherapy, chemotherapy or immunotherapy in our hospital
* Understand and fill in a variety of rating scales
* Informed consent, voluntary participation in this study

Exclusion Criteria:

* Neoadjuvant chemotherapy patients
* Intestinal obstruction or gastrointestinal bleeding
* Severe heart, lung and renal insufficiency
* Coagulopathy
* Clinical diagnosis with diabetes and other metabolic diseases
* The expected survival time is less than 1 month
* With cognitive dysfunction or poor coordination
* Allergy to creatine or curcumin
* With a history of drug abuse
* Doctors or researchers deem unsuitable for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
L3 skeletal muscle index(c㎡/㎡) | 0-month
  CT scans L3 cross-sectional skeletal muscle area/height²
L3 skeletal muscle index(c㎡/㎡) | 1-month
  CT scans L3 cross-sectional skeletal muscle area/height²
Appendicular skeletal muscle mass index(kg/㎡) | 0-month
  Appendicular skeletal muscle mass(ASM)is measured by bioelectrical impedance analysis(BIA), the ASM index (ASM/height²)is calculated.
Appendicular skeletal muscle mass index(kg/㎡) | 1-month
  Appendicular skeletal muscle mass(ASM)is measured by bioelectrical impedance analysis(BIA), the ASM index (ASM/height²)is calculated.

SECONDARY OUTCOMES:
Pre-albumin concentration(mg/L) | 0-month
  Serological pre-albumin concentration
Pre-albumin concentration(mg/L) | 1-month
  Serological pre-albumin concentration
Albumin concentration(g/L) | 0-month
  Serological albumin concentration
Albumin concentration(g/L) | 1-month
  Serological albumin concentration
Body Mass Index(kg/㎡) | 0-month
  body weight/height²
Body Mass Index(kg/㎡) | 1-month
  body weight/height²
Nutrition intake level(%) | 0-month
  Investigate the ratio of actual energy and protein intake levels to target intake levels
Nutrition intake level(%) | 1-month
  Investigate the ratio of actual energy and protein intake levels to target intake levels
PG-SGA score | 0-month
  Scored Patient-Generated Subjective Global Assessment(PG-SGA)：(0-1，stage A；2-8，stage B；≥9，stageC)
PG-SGA score | 1-month
  Scored Patient-Generated Subjective Global Assessment(PG-SGA)：(0-1，stage A；2-8，stage B；≥9，stageC)
Functional Assessment of Anorexia/Cachexia Therapy(FAACT) | 0-month
  Anorexia/Cachexia Sub-scale-12：score 0～24，Anorexia/Cachexia
Functional Assessment of Anorexia/Cachexia Therapy(FAACT) | 1-month
  Anorexia/Cachexia Sub-scale-12：score 0～24，Anorexia/Cachexia
Survival rate(%) | 1-month
  (Number of surviving cases after 1 month of follow-up)/(number of cases at the beginning of follow-up) ×100%
Survival rate(%) | 3-month
  (Number of surviving cases after 3 month of follow-up)/(number of cases at the beginning of follow-up) ×100%

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05856500/Prot_SAP_002.pdf
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05856500/ICF_003.pdf